CLINICAL TRIAL: NCT01498484
Title: A Phase II Study of the Therapeutic Effects Of Epstein-Barr Virus Immune T-Lymphocytes Derived From a Normal HLA-Compatible Or Partially-Matched Third-Party Donor in the Treatment of EBV Lymphoproliferative Disorders and EBV-Associated Malignancies
Brief Title: Therapeutic Effects of Epstein-Barr Virus Immune T-Lymphocytes Derived From a Normal HLA-Compatible Or Partially-Matched Third-Party Donor in the Treatment of EBV Lymphoproliferative Disorders and EBV-Associated Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Atara Biotherapeutics (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-130
Expanded Access: NCT02822495 (No longer available)
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Results first posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-09

CONDITIONS: EBV-induced Lymphomas; EBV-associated Malignancies; Transplant Patients With EBV Viremia at High Risk for Developing a Recurrent EBV Lymphoma
Keywords: EBV-specific T-cell lines; 11-130

ARMS (9):
- HCT EBV+ PTLD R/R Rituximab (Experimental): Patients with Epstein-Barr virus positive (EBV+) posttransplant lymphoproliferative disorders (PTLD) hematopoietic cell transplant (HCT) who were relapse/refractory (R/R) to rituximab will receive IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: EBV-specific T cells (EBV-CTLs)
- SOT EBV+ PTLD R/R Rituximab (Experimental): Patients with EBV+PTLD solid organ transplant (SOT) who were R/R to rituximab or R/R to rituximab and chemotherapy will receive IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After 3 week observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: EBV-specific T cells (EBV-CTLs)
- EBV+ AID-LPD (Experimental): Patients with EBV+ acquired immunodeficiency (AID) lymphoproliferative disorder (LPD) will receive IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity
  Interventions: Biological: EBV-specific T cells (EBV-CTLs)
- EBV+ PID-LPD (Experimental): Patients with EBV+ primary immunodeficiency (PID) LPD will receive IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: EBV-specific T cells (EBV-CTLs)
- EBV+ Viremia (Experimental): Patients with EBV+ viremia will receive IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: EBV-specific T cells (EBV-CTLs)
- EBV+ Leiomyosarcoma (Experimental): Patients with EBV+ leiomyosarcoma (LMS) will receive IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: EBV-specific T cells (EBV-CTLs)
- EBV+ Lymphoma (Experimental): Patients with EBV+ lymphoma will receive IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: EBV-specific T cells (EBV-CTLs)
- EBV+ NPC (Experimental): Patients with EBV+ nasopharyngeal carcinoma (NPC) will receive IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: EBV-specific T cells (EBV-CTLs)
- EBV+ Other Solid Tumor (Experimental): Patients with EBV+ other solid tumors will receive IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and will be observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: EBV-specific T cells (EBV-CTLs)

INTERVENTIONS:
Biological: EBV-specific T cells (EBV-CTLs) — EBV-CTLs are cytotoxic T lymphocytes that specifically kill cells presenting EBV protein antigens including EBV-transformed B lymphocytes responsible for EBV-associated lymphomas and lymphoproliferative disorders.
  Other Names: tabelecleucel; tab-cel®; ATA129

SUMMARY:
This is a Phase II trial to evaluate the efficacy and safety of human leukocyte antigen (HLA) partially-matched third-party allogeneic Epstein-Barr virus cytotoxic T lymphocytes (EBV-CTLs) for the treatment of EBV-induced lymphomas and EBV-associated malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented EBV antigen positive lymphoproliferative disease, lymphoma or other EBV-associated malignancy.

OR

* Evaluable disease as demonstrated by clinical and/or radiologic studies with current or prior elevated blood levels of EBV DNA exceeding 500 copies/ml by quantitative real time polymerase chain reaction (PCR).

OR

* Persistent or recurrent elevations in levels of EBV DNA exceeding 500 copies/ml in patients previously treated for EBV-LPD with chemotherapy and/or rituximab who do not yet have clinically or radiologically evaluable disease but are at high risk of disease recurrence.
* EBV-specific T cells are available for adoptive immune cell therapy from a consenting third party donor. The third party EBV-CTLs to be administered will be selected on the basis of two criteria: 1) that they are matched for at least 2 HLA antigens and 2) that they are restricted by an allele shared with the EBV+ malignancy (if known), or with the donor in HSCT recipients, or patient in organ transplant or immunodeficient patients
* KPS or Lansky score ≥ 20.
* A life expectancy of at least 6 weeks.
* Adequate bone marrow, heart, lung, liver and kidney function at the time of treatment with EBV-specificT cells is initiated, including:

  1. Absolute neutrophil count (ANC) ≥ 1,000/µL, with or without GCSF support
  2. Platelets ≥ 20,000/µL
  3. Creatinine ≤ 2.0mg/dl
  4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) < 3.0x and total bilirubin < 2.5x the institutional upper limit of normal (ULN)
  5. Stable blood pressure and circulation not requiring pressor support
  6. Adequate cardiac function as demonstrated by EKG and/or echocardiographic evidence (may be performed within 30 days prior to treatment)
* However, abnormalities of specific organs will not be considered grounds for exclusion if they are the result of the EBV+ malignancy or its treatment (e.g. a renal allograft recipient with an EBV LPD may be on dialysis because the allograft was rejected when the immune suppression was stopped as a first approach to treatment of the EBV LPD). At the discretion of the investigator, patients with elevated but stable creatinine will not be precluded from treatment on study.
* There is no age restriction to eligibility for this protocol.

It is expected that five types of patients afflicted with EBV-associated lymphomas, lymphoproliferative diseases or malignancies will be referred and will consent to participate in this trial. These are:

1. Patients developing EBV lymphomas or lymphoproliferative disorders following an allogeneic hematopoietic progenitor stem cell transplant (HSCT) (ie, marrow, PBSC, or umbilical cord blood).
2. Patients developing EBV lymphomas or lymphoproliferative disorders following an allogeneic organ transplant.
3. Patients with AIDS developing EBV lymphomas or lymphoproliferative diseases as a consequence of the profound acquired immunodeficiency induced by HIV.
4. Patients who develop EBV lymphomas or lymphoproliferative diseases or other EBV-associated malignancy as a consequence of profound immunodeficiencies associated with a congenital immune deficit or acquired as a sequela of anti-neoplastic or immunosuppressive therapy.
5. Patients who develop other EBV-associated malignancies without pre-existing immune deficiency, including: EBV+ Hodgkin's and Non-Hodgkin's disease, EBV+ nasopharyngeal carcinoma, EBV+ hemophagocytic lymphohistiocytosis, or EBV+ leiomyosarcoma.

Exclusion Criteria:

The following patients will be excluded from this study:

* Patients with active (grade 2-4) acute graft vs. host disease (GVHD), chronic GVHD or an overt autoimmune disease (e.g. hemolytic anemia) requiring high doses of glucocorticosteroid (>0.5 mg/kg/day prednisone or its equivalent) as treatment
* Patients who are pregnant
* Patients with severe comorbidities, not related to their EBV-associated malignancy, that would be expected to preclude their survival for the 6 weeks required to assess response of T cell therapy
* Patients eligible for MSK protocol #16-803 (EBV-CTL-201)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minoti Hiremath, MD, Study Director — Atara Biotherapeutics
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Prockop S, Doubrovina E, Suser S, Heller G, Barker J, Dahi P, Perales MA, Papadopoulos E, Sauter C, Castro-Malaspina H, Boulad F, Curran KJ, Giralt S, Gyurkocza B, Hsu KC, Jakubowski A, Hanash AM, Kernan NA, Kobos R, Koehne G, Landau H, Ponce D, Spitzer B, Young JW, Behr G, Dunphy M, Haque S, Teruya-Feldstein J, Arcila M, Moung C, Hsu S, Hasan A, O'Reilly RJ. Off-the-shelf EBV-specific T cell immunotherapy for rituximab-refractory EBV-associated lymphoma following transplantation. J Clin Invest. 2020 Feb 3;130(2):733-747. doi: 10.1172/JCI121127. PMID 31689242
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- HCT EBV+ PTLD R/R Rituximab: Participants with Epstein-Barr virus positive (EBV+) posttransplant lymphoproliferative disorders (PTLD) hematopoietic cell transplant (HCT) who were relapse/refractory (R/R) to rituximab received IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- SOT EBV+ PTLD R/R Rituximab: Participants with EBV+PTLD solid organ transplant (SOT) who were R/R to rituximab or R/R to rituximab and chemotherapy received IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and were observed for 3 weeks. After 3 week observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ AID-LPD: Participants with EBV+ acquired immunodeficiency (AID) lymphoproliferative disorder (LPD) received IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity. Results from participants in this arm are being excluded due to the low single digit numbers of participants; these low numbers pose a risk for participant re-identification in these rare indications in this single center study.
- EBV+ PID-LPD: Participants with EBV+ primary immunodeficiency (PID) LPD received IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity. Results from participants in this arm are being excluded due to the low single digit numbers of participants; these low numbers pose a risk for participant re-identification in these rare indications in this single center study.
- EBV+ Viremia: Participants with EBV+ viremia received IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity. Results from participants in this arm are being excluded due to the low single digit numbers of participants; these low numbers pose a risk for participant re-identification in these rare indications in this single center study.
- EBV+ Leiomyosarcoma: Participants with EBV+ leiomyosarcoma (LMS) received IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity. Results from participants in this arm are being excluded due to the low single digit numbers of participants; these low numbers pose a risk for participant re-identification in these rare indications in this single center study.
- EBV+ Lymphoma: Participants with EBV+ lymphoma received IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ NPC: Participants with EBV+ nasopharyngeal carcinoma (NPC) received IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ Other Solid Tumor: Participants with EBV+ other solid tumors received IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity. Results from participants in this arm are being excluded due to the low single digit numbers of participants; these low numbers pose a risk for participant re-identification in these rare indications in this single center study.
Period: Overall Study
Arm/Group | HCT EBV+ PTLD R/R Rituximab | SOT EBV+ PTLD R/R Rituximab | EBV+ AID-LPD | EBV+ PID-LPD | EBV+ Viremia | EBV+ Leiomyosarcoma | EBV+ Lymphoma | EBV+ NPC | EBV+ Other Solid Tumor
Started | 25 | 10 | 3 | 3 | 2 | 3 | 25 | 14 | 2
Completed | 11 | 3 | 1 | 0 | 1 | 2 | 3 | 0 | 0
Not Completed | 14 | 7 | 2 | 3 | 1 | 1 | 22 | 14 | 2
Not completed — Death | 6 | 3 | 1 | 1 | 0 | 0 | 10 | 1 | 0
Not completed — Physician Decision | 3 | 2 | 1 | 1 | 0 | 0 | 8 | 13 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 5 | 2 | 0 | 0 | 1 | 0 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least one dose of tabelecleucel. Results from arms with <= 3participants (EBV+ AID-LPD, EBV+ PID-LPD, EBV+ Viremia, EBV+ Leiomyosarcoma, and EBV+ Other Solid Tumor) are being excluded due to the low single digit numbers of participants; these low numbers pose a risk for participant re-identification in these rare indications in this single center study.
Groups:
- HCT EBV+ PTLD R/R Rituximab: Participants with EBV+ PTLD HCT who were R/R to rituximab received IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- SOT EBV+ PTLD R/R Rituximab: Participants with EBV+PTLD SOT who were R/R to rituximab or R/R to rituximab and chemotherapy received IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and were observed for 3 weeks. After 3 week observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- EBV+ NPC: Participants with EBV+ NPC received IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | HCT EBV+ PTLD R/R Rituximab | SOT EBV+ PTLD R/R Rituximab | EBV+ Lymphoma | EBV+ NPC | Total
Number analyzed (Participants) | 25 | 10 | 25 | 14 | 74
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 5 | 4 | 2 | 2 | 13
  >=18 years | 20 | 6 | 23 | 12 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 15 | 4 | 37
  Male | 14 | 3 | 10 | 10 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 4 | 0 | 3 | 3 | 10
  Unknown or Not Reported | 19 | 10 | 21 | 11 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 5 | 11 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 2 | 7
  White | 17 | 9 | 15 | 1 | 42
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The ORR is defined as percentage of participants with best overall response of complete remission/response (CR) or partial remission/response (PR) based on investigator's assessment. For participants with clinically and/or radiologically evident EBV LPD or malignancies, CR is complete resolution of all clinical and radiologic evidence of lymphoma, confirmed by biopsy of the affected tissues when indicated, lasting for at least 3 weeks following completion of a cycle of tabelecleucel; and PR is a 50 % or greater reduction in the size of all lymphomatous lesions as determined by computed tomography (CT) or magnetic resonance imaging (MRI) measurements of tumor volume, which was maintained for at least 3 weeks following completion of a cycle of tabelecleucel. For participants without clinically and/or radiologically evident tumors with increasing levels of EBV DNA, CR is clearance of EBV without subsequent development of EBV+ LPD; and PR is at least a 10-fold decrease in EBV DNA levels.
Time Frame: From Day 1 through 65.3 months after Day 1 dose
Population: Full analysis set included all participants who received at least one dose of tabelecleucel.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HCT EBV+ PTLD R/R Rituximab | SOT EBV+ PTLD R/R Rituximab | EBV+ Lymphoma | EBV+ NPC
Number analyzed (Participants) | 25 | 10 | 25 | 14
Percentage of participants | 68.0 [46.5 to 85.1] | 50.0 [18.7 to 81.3] | 16.0 [4.5 to 36.1] | 14.3 [1.8 to 42.8]

2. Secondary Outcome: Overall Survival (OS)
Description: The OS is defined as the time from the first dose of tabelecleucel to the date of death due to any cause. The OS was estimated using Kaplan-Meier method. Participants who were lost to follow-up or still alive were censored on the last known-to-be-alive date.
Time Frame: From Day 1 through 65.3 months after Day 1 dose
Population: Full analysis set included all participants who received at least one dose of tabelecleucel. Participants who were lost to follow-up or still alive were censored on the last known-to-be-alive date.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HCT EBV+ PTLD R/R Rituximab | SOT EBV+ PTLD R/R Rituximab | EBV+ Lymphoma | EBV+ NPC
Number analyzed (Participants) | 25 | 10 | 25 | 14
Months | NA [7.1 to NA] — Median and upper limit of confidence interval are not estimable due to insufficient events being observed at the time of the analysis. | 14.9 [0.4 to NA] — Upper limit of confidence interval is not estimable due to insufficient events being observed at the time of the analysis. | 12.3 [1.5 to 21.6] | NA [4.9 to NA] — Median and upper limit of confidence interval are not estimable due to insufficient events being observed at the time of the analysis.

3. Secondary Outcome: OS Rate at 12 Months
Description: Percentage of participants with OS at 12 months are reported. The OS is defined as the time from the first dose of tabelecleucel to the date of death due to any cause. The OS was estimated using Kaplan-Meier method. Participants who were lost to follow-up or still alive were censored on the last known-to-be-alive date.
Time Frame: From Day 1 through 12 months after Day 1 dose
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HCT EBV+ PTLD R/R Rituximab | SOT EBV+ PTLD R/R Rituximab | EBV+ Lymphoma | EBV+ NPC
Number analyzed (Participants) | 25 | 10 | 25 | 14
Percentage of participants | 68.0 [46.1 to 82.5] | 60.0 [25.3 to 82.7] | 50.3 [29.1 to 68.2] | 77.9 [45.9 to 92.3]

4. Secondary Outcome: OS Follow-up Time
Description: The OS follow-up time are reported. The OS is defined as the time from the first dose of tabelecleucel to the date of death due to any cause. The OS was estimated using Kaplan-Meier method. Participants who were lost to follow-up or still alive were censored on the last known-to-be-alive date.
Time Frame: From Day 1 through 65.3 months after Day 1 dose
Population: Full analysis set included all participants who received at least one dose of tabelecleucel.
Measure: Median (Full Range); unit: Months
Arm/Group | HCT EBV+ PTLD R/R Rituximab | SOT EBV+ PTLD R/R Rituximab | EBV+ Lymphoma | EBV+ NPC
Number analyzed (Participants) | 25 | 10 | 25 | 14
Months | 23.33 [0.6 to 60.6] | 14.88 [0.4 to 55.4] | 7.20 [0.3 to 65.3] | 16.0 [3.2 to 46.5]

5. Secondary Outcome: Time to Response (TTR)
Description: The TTR is defined as the time from the date of the first dose of tabelecleucel to the date of a PR or CR, whichever occurred first. For participants with clinically and/or radiologically evident EBV LPD or malignancies, CR is defined as complete resolution of all clinical and radiologic evidence of lymphoma, confirmed by biopsy of the affected tissues when indicated, lasting for at least 3 weeks following completion of a cycle of tabelecleucel; and a PR is defined as a 50 % or greater reduction in the size of all lymphomatous lesions as determined by CT or MRI scan measurements of tumor volume, which was maintained for at least 3 weeks following completion of a cycle of tabelecleucel. For participants without clinically and/or radiologically evident tumors with increasing levels of EBV DNA, CR is defined as clearance of EBV without subsequent development of EBV+ LPD; and PR is defined as at least a 10-fold decrease in EBV DNA levels.
Time Frame: From Day 1 through 65.3 months after Day 1 dose
Population: Full analysis set included all participants who received at least one dose of tabelecleucel. Participants who achieved CR or PR were analyzed for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | HCT EBV+ PTLD R/R Rituximab | SOT EBV+ PTLD R/R Rituximab | EBV+ Lymphoma | EBV+ NPC
Number analyzed (Participants) | 17 | 5 | 4 | 2
Months | 1.77 [0.7 to 6.4] | 3.32 [1.6 to 5.4] | 2.28 [1.2 to 8.4] | 1.76 [1.2 to 2.3]

ADVERSE EVENTS:
Time Frame: From Day 1 through 65.3 months after Day 1 dose
Description: Combined AE data for all enrolled participants are reported because few arms had <=3 participants which poses a risk of participant identification with rare indications in this study. Treatment-emergent SAEs includes events collected retrospectively and prospectively per protocol. Non-serious AEs were not collected, hence reported as '0'. In participant flow, 'Deaths' are reported as a reason for study discontinuation, whereas in 'All-Cause Mortality' deaths due to any cause are reported.
Groups:
- Overall Total: All eligible participants with EBV+ received IV infusion of tabelecleucel 2 × 10^6 T-cells/kg on Days 1, 8, and 15 and were observed for 3 weeks. After the observation period, additional courses (2 courses) may have been provided in the absence of disease progression or unacceptable toxicity.
Arm/Group | Overall Total
All-Cause Mortality (participants affected / at risk) | 46/87
Serious Adverse Events (participants affected / at risk) | 46/87
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Total (N=87)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (6)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis constrictive (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 13 (13)
Non-cardiac chest pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 8 (8)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 10 (13)
Otitis media (Infections and infestations) | 1 (1)
Periorbital infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 3 (3)
Skin infection (Infections and infestations) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 2 (3)
Encephalopathy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (4)
Mental status changes (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Embolism (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (3)

LIMITATIONS AND CAVEATS:
In this investigator-led study, scans were only collected as clinically indicated in lieu of a defined schedule; therefore, disease assessment endpoints (duration of response, durable response rate, progression-free survival, time to progression) may not be reliable, hence not reported. Study 11-130 was designed for patient treatment and conducted mostly as investigator-sponsored, single-center until Atara assumed responsibility, then relevant data was transferred from the investigator to Atara.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT01498484/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT01498484/SAP_001.pdf